CLINICAL TRIAL: NCT04346316
Title: A Randomized, Double Blind and Placebo-Controlled Phase II Study to Evaluate the Efficacy and Safety of SHR0302 Tablets in Adult Patients With Alopecia Areata
Brief Title: A Phase II Study in Patients With Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSJ10521
Record Dates: First submitted 2020-01-07; First posted 2020-04-15 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2020-11

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SHR0302 Dose#1 (Active Comparator)
  Interventions: Drug: SHR0302
- SHR0302 Dose#2 (Active Comparator)
  Interventions: Drug: SHR0302
- SHR0302 Dose#3 (Active Comparator)
  Interventions: Drug: SHR0302
- Placebo (Placebo Comparator)
  Interventions: Drug: SHR0302

INTERVENTIONS:
Drug: SHR0302 — Oral tablets taken once daily (QD)

SUMMARY:
This is a global Phase 2 study to evaluate the safety and effectiveness of an investigational study drug (called SHR0302) in adults with moderate to severe alopecia areata.

DETAILED DESCRIPTION:
The study is placebo-controlled, meaning that some patients entering the study will not receive active study drug but will receive tablets with no active ingredients (a placebo). This is a dose-ranging study, investigating 3 different dosing regimens. It will be double-blinded, meaning that the sponsor, the study doctors, the staff, and the patients will not know whether a patient is on active study drug (or the dose) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18-65 years of age (both inclusive), at the time of informed consent;
* Must have moderate to severe alopecia areata.

Exclusion Criteria:

* Other types of alopecia or other diseases that can cause hair loss
* Other scalp diseases that could interfere with assessment of hair loss/regrowth
* Any previous use of any Janus kinase (JAK) inhibitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in Severity of Alopecia Tool (SALT) score | week 24
  Severity of alopecia tool is a quantitative assessment of AA severity based on scalp hair loss

CONTACTS AND LOCATIONS:
Locations (31):
- United States (7):
  - Quest Dermatology Research, Northridge, California
  - Moore Clinical Research, Brandon, Florida
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - Skin Search of Rochester, Inc, Rochester, New York
  - Dermatologists of Southwest Ohio, Mason, Ohio
  - The Skin Wellness Center, Knoxville, Tennessee
  - Progressive Clinical Research, San Antonio, Texas
- Australia (6):
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - Novatrials, Kogarah, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Skin Health Institute, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Sinclair Dermatology, Melbourne, Victoria
- China (18):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Traditional Chinese medicine Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Dermatology Hospital of Nanfang Medical University, Guangzhou, Guangdong
  - The Dermatology Hospital of Nanfang Medical University, Guangzhou, Guangzhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jiangsu Province People's Hospital, Nanjin, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - SIR RUN RUN Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang